CLINICAL TRIAL: NCT06734104
Title: The Effect of an Interactive Video Developed for the Care of Surgical Patients Wearing Anti-Embolism Stockings on Nursing Students' Learning: A Randomized Controlled Experimental Study
Brief Title: The Effect of an Interactive Video on Nursing Students' Learning in the Care of Anti-Embolism Stockings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esra Cantürk (Other)
Responsible Party: Sponsor-Investigator, Esra Cantürk, PhD Student and Expert Nurse Esra Cantürk [ECanturk], Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 26.11.2024-E.1101844
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2024-12

CONDITIONS: Nursing Students; Nursing Education; Surgical Nursing
Keywords: anti-embolism stocking; interactive video; nursing students; nursing education; surgical nursing

STUDY DESIGN:
Intervention Model Description: This study protocol describes a single-center, randomized controlled parallel-group single-blind experimental study (1:1) to be conducted with nursing students at a public university in a province of Turkey. The protocol has been prepared in accordance with the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) guidelines. The sample will include 60 students, with 30 in the experimental group and 30 in the active control group. Data will be collected using the Student Demographic Characteristics Form, the Perioperative Anti-Embolism Stockings Care Knowledge Assessment Form, the Perioperative Anti-Embolism Stockings Application Skills Assessment Form, and the Interactive Video Evaluation Form, all of which were developed by the researchers based on the literature. The study will evaluate the impact of the interactive video developed for the care of surgical patients wearing anti-embolism stockings on the knowledge and skill levels of nursing students.
Who Masked: Participant, Outcomes Assessor
Masking Description: In the study, the researchers will be aware of the groups to which the students are assigned in order to plan the study. Since the students in the experimental group will receive an interactive video and those in the active control group will receive a non-interactive video, the students will not know their group assignment, ensuring participant blinding. Therefore, the study is single-blinded. During the process of obtaining informed consent, students will be informed that both groups will receive education on the subject through video. Additionally, students' skills will be assessed by three experts in the field of nursing, independent of the researchers. The evaluators will not be informed about the students' group assignments, ensuring blinding for the evaluators. Blinding will also be maintained during data analysis and reporting. Data entries will be coded as "A" and "B" without specifying whether they belong to the experimental or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Video Group (Experimental)
  Interventions: Other: Interactive Video Education
- Control : Non-Interactive Video Group (Active Comparator)
  Interventions: Other: Non-Interactive Video Education

INTERVENTIONS:
Other: Interactive Video Education — After participants are informed about the study, eligible individuals (based on inclusion and exclusion criteria) will be identified. From the students deemed eligible for the study group, 60 students will be selected using a simple random sampling method by an independent statistician. Informed consent will be obtained from students who agree to participate in the study. Initially, a pre-test will be administered to the 60 selected students. Following the pre-test, the students will be randomly assigned to the experimental and active control groups using a simple randomization method. The researcher will provide the interactive video to the students in the experimental group. After one week of interactive video training for the experimental group, a post-test will be administered to all students.
  Arms: Interactive Video Group
Other: Non-Interactive Video Education — After participants are informed about the study, eligible individuals (based on inclusion and exclusion criteria) will be identified. From the students deemed eligible for the study group, 60 students will be selected using a simple random sampling method by an independent statistician. Informed consent will be obtained from the students who agree to participate in the study. Initially, a pre-test will be administered to the 60 selected students. After the pre-test, the 60 students will be randomly assigned to the experimental and active control groups using a simple randomization method. The researcher will provide the non-interactive video to the students in the active control group. After one week of watching the non-interactive video, a post-test will be administered to all students.
  Arms: Control : Non-Interactive Video Group

SUMMARY:
This study will be conducted as a randomized controlled trial with a parallel design to determine the impact of an interactive video developed for the care of surgical patients wearing anti-embolism stockings on nursing students' learning outcomes. The research hypotheses are as follows:

H0a: There is no statistically significant difference in knowledge scores regarding anti-embolism stocking application between the intervention and control groups.

H0b: There is no statistically significant difference in knowledge scores regarding anti-embolism stocking application over time.

H0c: There is no statistically significant difference in skill scores regarding anti-embolism stocking application between the intervention and control groups.

H0d: There is no statistically significant difference in skill scores regarding anti-embolism stocking application over time.

H0e: There is no statistically significant difference in knowledge and skill scores regarding anti-embolism stocking application based on the interaction between group and time factors.

DETAILED DESCRIPTION:
The study will be conducted using a randomized controlled experimental design with third-year nursing students who have successfully completed their second year at a public university in a province of Turkey. The sample will include 60 students, with 30 in the experimental group and 30 in the active control group. Data will be collected using the Student Demographic Characteristics Form, the Perioperative Anti-Embolism Stockings Care Knowledge Assessment Form, the Perioperative Anti-Embolism Stockings Application Skills Assessment Form, and the Interactive Video Evaluation Form, all of which were developed by the researchers based on the literature. The study will evaluate the impact of the interactive video developed for the care of surgical patients wearing anti-embolism stockings on the knowledge and skill levels of nursing students.

ELIGIBILITY:
Inclusion Criteria:

* The student must own a smartphone, tablet, or laptop/desktop computer capable of downloading the video.
* The student must have internet access.
* The student must be willing to participate in the study voluntarily.

Exclusion Criteria:

* Graduates of health vocational high schools.
* Students who have failed the Surgical Diseases Nursing course.
* Students who have not participated in any of the stages of the study.
* Students who voluntarily decide to withdraw from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Knowledge level regarding perioperative anti-embolism stockings care | From enrollment to the end of intervention at 2 weeks
  Perioperative Anti-Embolism Stocking Care Knowledge Assessment Form consists of 18 multiple-choice questions. The researchers have developed the knowledge assessment questions regarding perioperative anti-embolism stockings care based on the literature. Each question has only one correct answer. Expert opinions were sought during the development of the knowledge assessment test to enhance content validity. The average item difficulty of the test was found to be 0.498. An ideal result would have an average item difficulty of 0.50. The average item discrimination index of the test was determined to be 0.431. A value higher than 0.35 indicates that the test has excellent discrimination power, meaning it is highly discriminative. The knowledge test will be scored on a scale of 100 points, with each correct answer worth 5.5 points. The minimum value is 0, and the maximum value is 99. A higher score indicates a better outcome.
Skill level regarding perioperative anti-embolism stockings care | From enrollment to the end of intervention at 2 weeks
  Perioperative Anti-Embolism Stocking Application Skills Assessment Form consists of 22 items. This form was developed by the researchers based on the literature. Expert opinions were sought during the development of the Skill Assessment Form to enhance content validity. In item number eight, the steps of neurovascular assessment are divided into seven sub-steps, and in item number 21, the situations to be recorded in the observation form for anti-embolism stockings are divided into four sub-categories. If a student fails to perform a skill, they will receive a score of zero (0), and if performed correctly, they will receive a score of one (1). The lowest score a student can receive is 0, and the highest score is 31. A higher score indicates a better outcome.

SECONDARY OUTCOMES:
The experimental group's opinions regarding the interactive video. | After the intervention is completed
  Interactive Video Evaluation Form on Perioperative Anti-Embolism Stocking Care includes a survey designed based on the literature to assess the opinions of students in the experimental group regarding the interactive video. In the first section of the form, students' positive and negative views about the interactive video game are explored through open-ended questions. The second section includes a total of 16 items, with 13 items related to the applicability of the interactive video game and three items related to its usability. Students will evaluate the game by assigning a score between one (1) and five (5) for each item. The minimum score is 16, and the maximum score is 80. A higher score indicates a better outcome. This form will be completed by the students in the experimental group after the final skill assessment is conducted.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Health Sciences, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided